CLINICAL TRIAL: NCT00903786
Title: A Long-term Extension Study of E2007 in Patients With Refractory Partial Seizures Uncontrolled With Other Anti-Epileptic Drugs (AEDs)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Eisai Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: E2007-J081-233
Record Dates: First submitted 2009-05-15; First posted 2009-05-18 (Estimated); Results first posted 2018-08-29 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2017-09

CONDITIONS: Refractory Partial Seizures
Keywords: Seizure; epilepsy
MeSH Terms: conditions — Seizures; Epilepsy | interventions — perampanel

ARMS (1):
- Perampanel (Experimental): Participants were treated with the perampanel dose that was administered in maintenance period of Study E2007-J081-231 (Study 231) [NCT00849212]. In some instances, a 1-step down-titration from the viewpoint of safety and up-titration to the maintenance dose of Study 231 was allowed. In general, 1 to 6 tablets of perampanel was administered orally as a 2-milligram (mg) tablet (2 mg to 12 mg) once daily before bedtime (under fed conditions as much as possible).
  The investigator, or subinvestigator, was allowed to complete the treatment by tapering the study drug after end of treatment or discontinuation (Follow-up Period), as appropriate. The taper period was 4 weeks at the longest.
  Interventions: Drug: perampanel

INTERVENTIONS:
Drug: perampanel — Patients will receive the same oral dosage (2 mg up to 12 mg once daily before bedtime) as used in the maintenance period of Study 231.
  Other Names: E2007; Fycompa

SUMMARY:
The purpose of this trial is to investigate the safety and tolerability of perampanel in long- term treatment in the patients with refractory partial epilepsy (uncontrolled with other anti-epileptic drugs) who completed Week 10 of Phase II Study E2007-J081-231 study.

ELIGIBILITY:
Inclusion criteria:

1. Patients who consent to the study entry on their free will before starting any trial-related activities.
2. Patients who participated in Study 231 and completed the required evaluation period (10 weeks).
3. Patients who are certainly and voluntarily able to participate in this study and record their seizures by themselves or have family members or caregivers (or nurses, if hospitalized) record the seizures. Patients who wish to continue perampanel treatment and necessitate receiving the long- term administration judged by the investigator or sub-investigator.

Exclusion criteria:

1. Pregnant or lactating women, women of child-bearing potential, women willing to become pregnant.
2. Patients who are ineligible judged by the investigator or sub investigator in light of medical history or complication at enrollment in treatment period.
3. Patients who operate heavy equipment or drive should not be recruited into the study.
4. Patients who are ineligible for study entry judged by the investigator or sub-investigator.

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2009-06-17 (Actual); Primary Completion 2016-08-08 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kazunori Saeki, Study Director — Neuroscience Clinical Development Section. JAC PCU. Eisai Co., Ltd.
Locations (9):
- Japan (9):
  - Kitakyushu, Fukuoka
  - Kobe, Hyōgo
  - Sendai, Miyagi
  - Komatsushimachō, Tokushima
  - Kodaira, Tokyo
  - Kyoto
  - Nagasaki
  - Niigata
  - Shizuoka

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Perampanel
Started | 21
Completed | 6
Not Completed | 15
Not completed — Physician Decision | 6
Not completed — Lack of Efficacy | 5
Not completed — Reason other than lack of efficacy | 4

BASELINE CHARACTERISTICS:
Population: The Safety Analysis Set (SAS) was defined as all participants who met the inclusion/exclusion criteria regarding "indication" (inclusion criteria number 5 of Study 231), who received at least one dose of study treatment, and who had at least one evaluable set of safety data.
Arm/Group | Perampanel
Number analyzed (Participants) | 21
Age, Continuous [Mean (Standard Deviation); unit: Years] | 36.5 (11.02)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 11

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs) and Serious Adverse Events (SAEs) as a Measure of Safety and Tolerability of Perampanel
Description: Safety was assessed by monitoring adverse events (AEs), adverse drug reactions, clinical laboratory parameters, vital signs, 12-lead electrocardiogram, and dependency questionnaire. AEs were graded on a 3-point scale; 1) mild: (Grade 1) discomfort noticed, but no disruption of normal daily activity, 2) moderate: (Grade 2) discomfort reduced or affected normal daily activity, and 3) severe: (Grade 3) incapacitating, with inability to work or to perform normal daily activity. AE severity associated with abnormal changes in laboratory parameters was assessed using the Ministry of Health and Welfare Notification Number 80 "Classification of Severity of Adverse Drug Reactions of Medicinal Products". TEAEs were defined as AEs that emerged during treatment (absent at pretreatment [Baseline]), reemerged during treatment (were present at pretreatment but stopped before treatment), or worsened in severity during treatment relative to the pretreatment state, when the AE was continuous.
Time Frame: From date of first dose up to 30 days after the last dose of study treatment, up to approximately 7 years 2 months
Population: as for baseline characteristics
Measure: Number; unit: Participants
Arm/Group | Perampanel
Number analyzed (Participants) | 21
Participants
  TEAEs | 21
  Treatment-related TEAEs | 11
  Serious TEAEs | 5
  TEAEs Leading to Study Treatment Dose Reduction | 2

2. Secondary Outcome: Percent Change in Total Seizure Frequency Per 28 Days for the Treatment Period Summarized Until Week 316
Description: Seizure frequency was derived from information (seizure count and type) recorded in the participant diary. The seizure frequency per 28 days was calculated as the number of seizures over the time interval multiplied by 28 and divided by the number of days in the interval. The percent change in 28-day seizure frequency from baseline was assessed for overall seizures, overall partial seizures, overall generalized seizures, and unclassified seizures. Of the 21 participants, 20 participants concomitantly used at least 1 inducer anti-epileptic drug (AED) (carbamazepine, phenytoin, phenobarbital, or primidone), and 1 participant used only non-inducer AEDs. The data is presented as median percent change with full range.
Time Frame: From Week 1 through Week 316 and Follow-up Period of the Extension Study, up to approximately 7 years 2 months
Population: The Efficacy Analysis Population (identical to the SAS for this study) was defined as all participants who met the inclusion/exclusion criteria regarding "indication" (inclusion criteria number 5 of Study 231), who received at least one dose of study treatment, and who had at least one data on efficacy.
Measure: Median (Full Range); unit: Percent change in seizure frequency
Groups:
- Perampanel: Participants were treated with the perampanel dose that was administered in maintenance period of Study E2007-J081-231 (Study 231) [NCT00849212]. In some instances, a 1-step down-titration from the viewpoint of safety and up-titration to the maintenance dose of Study 231 was allowed. In general, 1 to 6 tablets of perampanel was administered orally as a 2-mg tablet (2 mg to 12 mg) once daily before bedtime (under fed conditions as much as possible).
  The investigator, or subinvestigator, was allowed to complete the treatment by tapering the study drug after end of treatment or discontinuation (Follow-up Period), as appropriate. The taper period was 4 weeks at the longest.
Arm/Group | Perampanel
Number analyzed (Participants) | 21
Percent change in seizure frequency
  Weeks 1 to 4 | -33.33 [-100.0 to 24.4]
  Weeks 5 to 8 | -36.36 [-100.0 to 38.9]
  Weeks 9 to 16 | -26.32 [-100.0 to 31.3]
  Weeks 17 to 28: number analyzed (Participants) | 20
  Weeks 17 to 28 | -36.67 [-100.0 to 15.3]
  Weeks 29 to 40: number analyzed (Participants) | 18
  Weeks 29 to 40 | -31.10 [-100.0 to 33.3]
  Weeks 41 to 52: number analyzed (Participants) | 17
  Weeks 41 to 52 | -49.36 [-100.0 to 5.0]
  Weeks 53 to 64: number analyzed (Participants) | 17
  Weeks 53 to 64 | -42.43 [-100.0 to 49.7]
  Weeks 65 to 76: number analyzed (Participants) | 17
  Weeks 65 to 76 | -36.09 [-100.0 to -1.2]
  Weeks 77 to 88: number analyzed (Participants) | 16
  Weeks 77 to 88 | -38.82 [-100.0 to 9.8]
  Weeks 89 to 100: number analyzed (Participants) | 16
  Weeks 89 to 100 | -57.65 [-100.0 to -9.9]
  Weeks 101 to 112: number analyzed (Participants) | 16
  Weeks 101 to 112 | -52.45 [-100.0 to 12.5]
  Weeks 113 to 124: number analyzed (Participants) | 16
  Weeks 113 to 124 | -57.49 [-100.0 to 28.2]
  Weeks 125 to 136: number analyzed (Participants) | 15
  Weeks 125 to 136 | -36.27 [-100.0 to 94.4]
  Weeks 137 to 148: number analyzed (Participants) | 13
  Weeks 137 to 148 | -41.81 [-100.0 to 23.1]
  Weeks 149 to 160: number analyzed (Participants) | 12
  Weeks 149 to 160 | -41.13 [-100.0 to -5.1]
  Weeks 161 to 172: number analyzed (Participants) | 10
  Weeks 161 to 172 | -39.76 [-100.0 to 68.9]
  Weeks 173 to 184: number analyzed (Participants) | 10
  Weeks 173 to 184 | -34.52 [-100.0 to 29.2]
  Weeks 185 to 196: number analyzed (Participants) | 9
  Weeks 185 to 196 | -34.12 [-100.0 to 64.1]
  Weeks 197 to 208: number analyzed (Participants) | 9
  Weeks 197 to 208 | -83.53 [-100.0 to 22.5]
  Weeks 209 to 220: number analyzed (Participants) | 9
  Weeks 209 to 220 | -58.97 [-100.0 to 53.3]
  Weeks 221 to 232: number analyzed (Participants) | 9
  Weeks 221 to 232 | -41.83 [-100.0 to 86.7]
  Weeks 233 to 244: number analyzed (Participants) | 7
  Weeks 233 to 244 | -75.29 [-100.0 to -26.5]
  Weeks 245 to 256: number analyzed (Participants) | 7
  Weeks 245 to 256 | -83.53 [-100.0 to -2.0]
  Weeks 257 to 268: number analyzed (Participants) | 7
  Weeks 257 to 268 | -83.53 [-100.0 to 58.5]
  Weeks 269 to 280: number analyzed (Participants) | 6
  Weeks 269 to 280 | -95.88 [-100.0 to 19.2]
  Weeks 281 to 292: number analyzed (Participants) | 6
  Weeks 281 to 292 | -83.35 [-100.0 to -26.5]
  Weeks 293 to 304: number analyzed (Participants) | 6
  Weeks 293 to 304 | -87.65 [-100.0 to -5.0]
  Weeks 305 to 316: number analyzed (Participants) | 3
  Weeks 305 to 316 | -99.59 [-100.0 to -75.3]
  Follow-up period: number analyzed (Participants) | 15
  Follow-up period | -8.40 [-74.5 to 230.9]

3. Secondary Outcome: Responder Rate During the Treatment Period-LOCF
Description: Responder rate (percentage of participants with greater than or equal to 50% reduction in seizure frequency for 28 days in the Treatment Period relative to that for 28 days in the observation period of Study 231 [responder]. If the reduction in seizure frequency is less than 50%, then the participants are considered as non-responders.
  LOCF = Last Observation Carried Forward.
Time Frame: Week 1 through Week 316 and Follow-up period of the Extension study, up to approximately 7 years 2 months
Population: Efficacy Analysis Population
Measure: Number; unit: Percentage of participants
Arm/Group | Perampanel
Number analyzed (Participants) | 21
Percentage of participants
  Weeks 1 to 4; Responder | 42.9
  Weeks 1 to 4; Non-Responder | 57.1
  Weeks 5 to 9; Responder | 42.9
  Weeks 5 to 9; Non-Responder | 57.1
  Weeks 9 to 16; Responder | 28.6
  Weeks 9 to 16; Non-Responder | 71.4
  Weeks 17 to 28; Responder: number analyzed (Participants) | 20
  Weeks 17 to 28; Responder | 40.0
  Weeks 17 to 28; Non-Responder: number analyzed (Participants) | 20
  Weeks 17 to 28; Non-Responder | 60.0
  Weeks 29 to 40; Responder: number analyzed (Participants) | 18
  Weeks 29 to 40; Responder | 44.4
  Weeks 29 to 40; Non-Responder: number analyzed (Participants) | 18
  Weeks 29 to 40; Non-Responder | 55.6
  Weeks 41 to 52; Responder: number analyzed (Participants) | 17
  Weeks 41 to 52; Responder | 47.1
  Weeks 41 to 52; Non-Responder: number analyzed (Participants) | 17
  Weeks 41 to 52; Non-Responder | 52.9
  Weeks 53 to 64; Responder: number analyzed (Participants) | 17
  Weeks 53 to 64; Responder | 41.2
  Weeks 53 to 64; Non-Responder: number analyzed (Participants) | 17
  Weeks 53 to 64; Non-Responder | 58.8
  Weeks 65 to 76; Responder: number analyzed (Participants) | 17
  Weeks 65 to 76; Responder | 41.2
  Weeks 65 to 76; Non-Responder: number analyzed (Participants) | 17
  Weeks 65 to 76; Non-Responder | 58.8
  Weeks 77 to 88; Responder: number analyzed (Participants) | 16
  Weeks 77 to 88; Responder | 31.3
  Weeks 77 to 88; Non-Responder: number analyzed (Participants) | 16
  Weeks 77 to 88; Non-Responder | 68.8
  Weeks 89 to 100; Responder: number analyzed (Participants) | 16
  Weeks 89 to 100; Responder | 56.3
  Weeks 89 to 100; Non-Responder: number analyzed (Participants) | 16
  Weeks 89 to 100; Non-Responder | 43.8
  Weeks 101 to 112; Responder: number analyzed (Participants) | 16
  Weeks 101 to 112; Responder | 50.0
  Weeks 101 to 112; Non-Responder: number analyzed (Participants) | 16
  Weeks 101 to 112; Non-Responder | 50.0
  Weeks 113 to 124; Responder: number analyzed (Participants) | 16
  Weeks 113 to 124; Responder | 56.3
  Weeks 113 to 124; Non-Responder: number analyzed (Participants) | 16
  Weeks 113 to 124; Non-Responder | 43.8
  Weeks 125 to 136; Responder: number analyzed (Participants) | 15
  Weeks 125 to 136; Responder | 40.0
  Weeks 125 to 136; Non-Responder: number analyzed (Participants) | 15
  Weeks 125 to 136; Non-Responder | 60.0
  Weeks 137 to 148; Responder: number analyzed (Participants) | 13
  Weeks 137 to 148; Responder | 38.5
  Weeks 137 to 148; Non-Responder: number analyzed (Participants) | 13
  Weeks 137 to 148; Non-Responder | 61.5
  Weeks 149 to 160; Responder: number analyzed (Participants) | 12
  Weeks 149 to 160; Responder | 50.0
  Weeks 149 to 160; Non- Responder: number analyzed (Participants) | 12
  Weeks 149 to 160; Non- Responder | 50.0
  Weeks 161 to 172; Responder: number analyzed (Participants) | 10
  Weeks 161 to 172; Responder | 40.0
  Weeks 161 to 172; Non-Responder: number analyzed (Participants) | 10
  Weeks 161 to 172; Non-Responder | 60.0
  Weeks 173 to 184; Responder: number analyzed (Participants) | 10
  Weeks 173 to 184; Responder | 40.0
  Weeks 173 to 184; Non-Responder: number analyzed (Participants) | 10
  Weeks 173 to 184; Non-Responder | 60.0
  Weeks 185 to 196; Responder: number analyzed (Participants) | 9
  Weeks 185 to 196; Responder | 44.4
  Weeks 185 to 196; Non-Responder: number analyzed (Participants) | 9
  Weeks 185 to 196; Non-Responder | 55.6
  Weeks 197 to 208; Responder: number analyzed (Participants) | 9
  Weeks 197 to 208; Responder | 66.7
  Weeks 197 to 208; Non-Responder: number analyzed (Participants) | 9
  Weeks 197 to 208; Non-Responder | 33.3
  Weeks 209 to 220; Responder: number analyzed (Participants) | 9
  Weeks 209 to 220; Responder | 55.6
  Weeks 209 to 220; Non-Responder: number analyzed (Participants) | 9
  Weeks 209 to 220; Non-Responder | 44.4
  Weeks 221 to 232; Responder: number analyzed (Participants) | 9
  Weeks 221 to 232; Responder | 44.4
  Weeks 221 to 232; Non-Responder: number analyzed (Participants) | 9
  Weeks 221 to 232; Non-Responder | 55.6
  Weeks 233 to 244; Responder: number analyzed (Participants) | 7
  Weeks 233 to 244; Responder | 57.1
  Weeks 233 to 244; Non-Responder: number analyzed (Participants) | 7
  Weeks 233 to 244; Non-Responder | 42.9
  Weeks 245 to 256; Responder: number analyzed (Participants) | 7
  Weeks 245 to 256; Responder | 85.7
  Weeks 245 to 256; Non-Responder: number analyzed (Participants) | 7
  Weeks 245 to 256; Non-Responder | 14.3
  Weeks 257 to 268; Responder: number analyzed (Participants) | 7
  Weeks 257 to 268; Responder | 85.7
  Weeks 257 to 268; Non-Responder: number analyzed (Participants) | 7
  Weeks 257 to 268; Non-Responder | 14.3
  Weeks 269 to 280; Responder: number analyzed (Participants) | 6
  Weeks 269 to 280; Responder | 83.3
  Weeks 269-280; Non-Responder: number analyzed (Participants) | 6
  Weeks 269-280; Non-Responder | 16.7
  Weeks 281 to 292; Responder: number analyzed (Participants) | 6
  Weeks 281 to 292; Responder | 83.3
  Weeks 281 to 292; Non-Responder: number analyzed (Participants) | 6
  Weeks 281 to 292; Non-Responder | 16.7
  Weeks 293 to 304; Responder: number analyzed (Participants) | 6
  Weeks 293 to 304; Responder | 83.3
  Weeks 293 to 304; Non-Responder: number analyzed (Participants) | 6
  Weeks 293 to 304; Non-Responder | 16.7
  Weeks 305 to 316; Responder: number analyzed (Participants) | 3
  Weeks 305 to 316; Responder | 100.0
  Weeks 305 to 316; Non-Responder: number analyzed (Participants) | 3
  Weeks 305 to 316; Non-Responder | 0.0
  Follow-up period; Responder: number analyzed (Participants) | 15
  Follow-up period; Responder | 20.0
  Follow-up period; Non-responder: number analyzed (Participants) | 15
  Follow-up period; Non-responder | 80.0

4. Secondary Outcome: The Patient Global Impression of Change (PGIC) at Week 52 and End of Treatment
Description: Each participant evaluated him/herself for PGIC at Week 52 of the Treatment Period and at the end of treatment (or discontinuation) by comparing seizure conditions during 4 weeks before Week 52 of the Treatment Period and those during 4 weeks before end of treatment (or discontinuation) of the open label extension study with those during 4 weeks before start of the Treatment Period of Study 231. Assessment was implemented based on frequency of seizure, severity of seizures, AEs, and overall conditions using the 7-grade scores. The evaluation used a 7-point scale with the scores 1: Very much improved, 2: Much improved, 3: Minimally improved, 4: No change, 5: Minimally worse, 6: Much worse, 7: Very much worse.
Time Frame: Week 52 and End of Treatment; up to approximately 7 years 2 months
Population: Efficacy Analysis Population
Measure: Number; unit: Percentage of participants
Arm/Group | Perampanel
Number analyzed (Participants) | 21
Percentage of participants
  Very much improved; Week 52: number analyzed (Participants) | 17
  Very much improved; Week 52 | 17.6
  Much improved; Week 52: number analyzed (Participants) | 17
  Much improved; Week 52 | 17.6
  Minimally improved; Week 52: number analyzed (Participants) | 17
  Minimally improved; Week 52 | 52.9
  No change; Week 52: number analyzed (Participants) | 17
  No change; Week 52 | 11.8
  Minimally worse; Week 52: number analyzed (Participants) | 17
  Minimally worse; Week 52 | 0.0
  Much worse; Week 52: number analyzed (Participants) | 17
  Much worse; Week 52 | 0.0
  Very much worse; Week 52: number analyzed (Participants) | 17
  Very much worse; Week 52 | 0.0
  Very much improved; End of Treatment | 14.3
  Much improved; End of Treatment | 14.3
  Minimally improved; End of Treatment | 28.6
  No change; End of Treatment | 38.1
  Minimally worse; End of Treatment | 4.8
  Much worse; End of Treatment | 0.0
  Very much worse; End of Treatment | 0.0

5. Secondary Outcome: The Clinical Global Impression of Change (CGIC) at Week 52 and End of Treatment
Description: The investigator evaluated each participant for CGIC at Week 52 of the Treatment Period and at the end of treatment (or discontinuation) by comparing medical conditions during 4 weeks before Week 52 of the Treatment Period and those during 4 weeks before end of treatment (or discontinuation) of the open label extension study with those during 4 weeks before start of the Treatment Period of Study 231. Assessment was implemented based on frequency of seizure, severity of seizures, AEs, and overall conditions using the 7-grade scores. The evaluation used a 7-point scale with the scores 1: Very much improved, 2: Much improved, 3: Minimally improved, 4: No change, 5: Minimally worse, 6: Much worse, 7: Very much worse.
Time Frame: Week 52 and End of Treatment, up to approximately 7 years 2 months
Population: Efficacy Analysis Population
Measure: Number; unit: Percentage of participants
Arm/Group | Perampanel
Number analyzed (Participants) | 21
Percentage of participants
  Very much improved; Week 52: number analyzed (Participants) | 17
  Very much improved; Week 52 | 11.8
  Much improved; Week 52: number analyzed (Participants) | 17
  Much improved; Week 52 | 5.9
  Minimally improved; Week 52: number analyzed (Participants) | 17
  Minimally improved; Week 52 | 64.7
  No change; Week 52: number analyzed (Participants) | 17
  No change; Week 52 | 17.6
  Minimally worse; Week 52: number analyzed (Participants) | 17
  Minimally worse; Week 52 | 0.0
  Much worse; Week 52: number analyzed (Participants) | 17
  Much worse; Week 52 | 0.0
  Very much worse; Week 52: number analyzed (Participants) | 17
  Very much worse; Week 52 | 0.0
  Very much improved; End of Treatment | 9.5
  Much improved; End of Treatment | 9.5
  Minimally improved; End of Treatment | 19.0
  No change; End of Treatment | 61.9
  Minimally worse; End of Treatment | 0.0
  Much worse; End of Treatment | 0.0
  Very much worse; End of Treatment | 0.0

ADVERSE EVENTS:
Time Frame: From date of first dose up to 30 days after the last dose of study treatment, up to approximately 7 years 2 months
Description: Treatment-emergent adverse events were defined as adverse events (AE) that started on or after the date and time of administration of first dose of test drug, but not later than 30 days after discontinuation from the study, or if the AE was present prior to the administration of the first dose of test drug, worsened in severity. AE severity was graded using Ministry of Health and Welfare Notification Number 80 Classification of Severity of Adverse Drug Reactions of Medicinal Products.
Arm/Group | Perampanel
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 5/21
Other Adverse Events (participants affected / at risk) | 21/21
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (N=21)
Pneumonia bacterial (Infections and infestations) | 1
Epilepsy (Nervous system disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Perampanel (N=21)
Nasopharyngitis (Infections and infestations) | 14
Gingivitis (Infections and infestations) | 2
Influenza (Infections and infestations) | 2
Gastroenteritis (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 1
Hordeolum (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Urinary tract infection (Infections and infestations) | 1
Pneumonia bacterial (Infections and infestations) | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1
Hyperuricaemia (Metabolism and nutrition disorders) | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 1
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Mental status changes (Psychiatric disorders) | 1
Dizziness (Nervous system disorders) | 6
Somnolence (Nervous system disorders) | 6
Headache (Nervous system disorders) | 4
Tremor (Nervous system disorders) | 2
Ataxia (Nervous system disorders) | 1
Epilepsy (Nervous system disorders) | 1
Partial seizures with secondary generalisation (Nervous system disorders) | 1
Conjunctivitis (Eye disorders) | 1
Diplopia (Eye disorders) | 1
Presbyopia (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 1
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 2
Gastritis (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Stomatitis (Gastrointestinal disorders) | 2
Abdominal pain upper (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric ulcer (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 1
Mouth haemorrhage (Gastrointestinal disorders) | 1
Oesophagitis (Gastrointestinal disorders) | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1
Acne (Skin and subcutaneous tissue disorders) | 2
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Drug eruption (Skin and subcutaneous tissue disorders) | 1
Eczema (Skin and subcutaneous tissue disorders) | 1
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 1
Hypohidrosis (Skin and subcutaneous tissue disorders) | 1
Skin fissures (Skin and subcutaneous tissue disorders) | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Arthritis (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1
Tenosynovitis (Musculoskeletal and connective tissue disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Prostatitis (Reproductive system and breast disorders) | 1
Malaise (General disorders) | 3
Pyrexia (General disorders) | 3
Irritability (General disorders) | 2
Feeling abnormal (General disorders) | 1
Feeling drunk (General disorders) | 1
Local swelling (General disorders) | 1
Thirst (General disorders) | 1
Gamma-glutamyltransferase increased (Investigations) | 3
Blood glucose increased (Investigations) | 2
Blood calcium decreased (Investigations) | 1
Blood creatine phosphokinase increased (Investigations) | 1
Blood creatinine increased (Investigations) | 1
Blood glucose decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Eosinophil count increased (Investigations) | 1
Glucose urine present (Investigations) | 1
Protein urine present (Investigations) | 1
Human chorionic gonadotropin increased (Investigations) | 1
Contusion (Injury, poisoning and procedural complications) | 12
Laceration (Injury, poisoning and procedural complications) | 4
Fall (Injury, poisoning and procedural complications) | 2
Rib fracture (Injury, poisoning and procedural complications) | 2
Mouth injury (Injury, poisoning and procedural complications) | 2
Excoriation (Injury, poisoning and procedural complications) | 2
Chillblains (Injury, poisoning and procedural complications) | 1
Foot fracture (Injury, poisoning and procedural complications) | 1
Hand fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Ligament sprain (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Thermal burn (Injury, poisoning and procedural complications) | 1
Tongue injury (Injury, poisoning and procedural complications) | 1
Ligament injury (Injury, poisoning and procedural complications) | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other